CLINICAL TRIAL: NCT03283293
Title: Study on Delineation of the Target Volumes and Determination of the Irradiation Doses in Untreated Nasopharyngeal Carcinoma (NPC) Treated With Intensity Modulated Radiation Therapy (IMRT)
Brief Title: Target Volume Delineation After NACT in LA-NPCarcinoma Patients Treated With NACT+ CCRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhao Chong, MD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTV Delineation after NACT
Record Dates: First submitted 2017-09-11; First posted 2017-09-14 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Neoadjuvant Chemotherapy; Intensity-modulated Radiation Therapy; Target Volume Delineation; Locoregional Failure Pattern; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Target volume delineation after NACT (Experimental)
  Interventions: Radiation: Target Volume Delineation after NACT

INTERVENTIONS:
Radiation: Target Volume Delineation after NACT — The gross tumor volumes of the primary site and the neck nodes (GTVnx and GTVnd) were delineated in accordance with the head and neck magnetic resonance imaging (MRI) and endoscopy, which obtained two weeks after the last cycle of NACT. The first clinical target volume (CTV1) was defined as the GTVnx plus a 5-10mm margin (2 to 3mm margin posteriorly) to encompass the high-risk sites of microscopic extension, the whole nasopharynx, and the location and extent of the primary tumor before NACT. The second clinical target volume (CTV2) was defined as the CTV1 plus a 5-10mm margin (2 to 3mm margin posteriorly) to encompass the low-risk sites of microscopic extension, the level of the lymph node located before NACT, and the elective neck area. The prescribed dose to GTVnx, GTVnd, CTV1 and CTV2 were 68Gy/30f, 62-66Gy/30f, 60Gy/30f and 54Gy/30f, respectively.

SUMMARY:
The gross tumor volumes of the primary site and the neck nodes (GTVnx and GTVnd) could be delineated according to the post-NACT tumor position and receive radical radiation dose, while the tumor disappear after NACT could be encompassed in the first clinical target volume (CTV1) and receive high preventive radiation dose. Through this method,it is more likely to achieve the ultimate goal that maximize the chance of cure while minimize the injury of surrounding normal tissues, maintaining organ function and life quality. Therefore, this stage II clinical trial was designed to study the prognosis and locoregional failure patterns of this target volume delineation method in LA-NPC treated with NACT plus CCRT.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed NPC;
2. no evidence of distant metastasis;
3. no previous treatment for NPC;
4. stages III-IVb disease according to the staging system of the 6th AJCC/UICC;
5. adequate liver, renal and bone marrow function;
6. Karnofsky Performance Status (KPS) ≥80 scores.

Exclusion Criteria:

1. fine-needle aspiration biopsy, incisional or excisional biopsy of neck lymph node, or neck dissection prior NACT;
2. disease progression during NACT;
3. presence of distant metastasis;
4. pregnancy or lactation;
5. previous malignancy or other concomitant malignant disease.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2001-02 (Actual); Primary Completion 2007-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
5-year loco-regional recurrence free survival (LRRFS) | Five years

SECONDARY OUTCOMES:
5-year local recurrence free survival (LRFS) | Five years
5-year regional recurrence free survival (RRFS) | Five years
5-year distant metastasis free survival (DMFS) | Five years
5-year disease specific survival (DSS) | Five years
5-year overall survival (OS) | Five years
Locoregional failure patterns | Five years
  The failures were categorized as occurring inside or outside the high dose target volume, depending on the location of Vrecur: "in field" if 95% of Vrecur was within the 95% isodose; "marginal" if 20% to 95% of Vrecur was within the 95% isodose, or "outside" if less than 20% of Vrecur was inside the 95% isodose.
Late toxicities | Five years
  The late toxicities were graded according to the Radiation Therapy Oncology Group radiation morbidity scoring criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Chong Zhao, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China